CLINICAL TRIAL: NCT06669520
Title: Correlation of Blood Serum Renalase and Microcirculation Obstruction in Patients with Acute Myocardial Infarction After Primary Percutaneous Coronary Intervention
Status: Recruiting | Type: Observational
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: K 24655
Record Dates: First submitted 2024-10-29; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This research will explore the association between blood serum renalase and microcirculation obstruction in patients with acute myocardial infarction (AMI) after primary percutaneous coronary intervention (PCI). The investigators aim to identify potential risk factors for microcirculation obstruction in AMI patients after PPCI.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. STEMI symptom onset time < 12 hours;
3. STEMI symptom onset time 12-48 hours with persistent ischemic symptoms, hemodynamic instability, or life-threatening ventricular arrhythmias;
4. High-risk NSTEMI;
5. Emergency PCI;
6. Voluntary informed consent.

Exclusion Criteria:

1. Non-obstructive acute myocardial infarction;
2. Severe chronic kidney disease (defined as estimated glomerular filtration rate < 20 mL/min per 1.73 m²);
3. Life expectancy < 1 year;
4. Pregnant or planning to become pregnant;
5. Emergency PCI failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include 200 patients diagnosed with acute myocardial infarction (AMI) who will undergo primary percutaneous coronary intervention (PCI) at the Third Xiangya Hospital of Central South University, from August 2024 to August 2025.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Microvascular Obstruction Assessed by Contrast-Enhanced Magnetic Resonance Imaging 3-7 Days After Percutaneous Coronary Intervention. | 3-7 days after PPCI
  Microvascular obstruction (MVO) was qualitatively recognized as a subendocardial lack of enhancement at first-pass perfusion (FPP) sequences and as a hypointense region within the hyperintense infarcted area at early gadolinium enhancement (EGE) and late gadolinium enhancement (LGE) sequences.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen Y, Li R, Fu R, Zhao L, Sheng Z, Xu K, Liu J, Huang W, Wen J, Zeng L, Ou Z, Jiang Z, Liu Y, Wang Y, Jiang W, Li X. Association between periprocedural change in serum renalase and microvascular obstruction in patients with STEMI after primary percutaneous coronary intervention: protocol for the ReMVOS prospective cohort study. BMJ Open. 2025 Nov 28;15(11):e110045. doi: 10.1136/bmjopen-2025-110045. PMID 41314850